CLINICAL TRIAL: NCT06870123
Title: A Prospective Randomized Clinical Study Evaluating the Outcomes of MINIMA Stem with DELTA TT or DELTA ST-C Cup After Total Hip Arthroplasty
Brief Title: Randomized MINIMA Stem with DELTA TT or DELTA ST-C
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-41
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minima Stem with ST-c Cup (Other): Minima Stem with ST-c Cup
  Interventions: Device: TT cup and ST-C cup
- Minima Stem with TT Cup (Other): Minima Stem with TT Cup
  Interventions: Device: TT cup and ST-C cup

INTERVENTIONS:
Device: TT cup and ST-C cup — Patients are allocated in 2 different group (one with ST-C Cup and another one with TT Cup)

SUMMARY:
This study is aimed to provide a clinical and radiographic evaluation of 120 suitable subjects who underwent a total hip arthroplasty with MINIMA stem coupled with Delta TT or Delta ST-C cup.

DETAILED DESCRIPTION:
This is a post-market, interventional, prospective, randomized, not comparative, open label study designed to reflect real life clinical practice as closely as possible.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Any race
* A diagnosis in the target hip of one or more of the following: a) non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis; b) rheumatoid arthritis; c) post-traumatic arthritis; d) fractures of femoral neck;
* patien willingness to partecipate and signature of informed consent form

Exclusion Criteria:

* local or systemic infection
* septicaemia
* persistent acute or chronic osteomyelitis
* confirmed nerve or muscle lesion compromising hip joint function
* vascular or nerve disease affecting the concerned limb
* poor bone stock (for example due to osteoporosis) compromising the stability of the implant
* metabolic disorders which may impair fixation and stability of the implant
* any concomitant disease and dependence that might affect the implanted prosthsis
* metal hypersensitivity to implant materials
* required revision of previous standard femoral stem
* women of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remail on an acceptable method of birth control throughout the entire study period
* life expectancy less than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score (HHS) | 3 years
  Functional changes in Harris Hip Score (HHS) from preoperative (baseline) to 3 years after surgery

SECONDARY OUTCOMES:
Harris Hip Score (HHS) | 5 years
  Functional changes in Harris Hip Score (HHS) from preoperative (baseline) to 5 years after surgery
Implant stability | 6 months, 1 year, 3 years, 5 years after surgery
  Radiographic implant evaluation and stability assessment at 6 months, 1 year, 3 years, 5 years after surgery
Oxford Hip Score (OHS) | 5 years
  Functional changes in Oxford Hip Score (OHS) from preoperative (baseline) to 5 years after surgery
Forgotten Joint Score (FJS) | 3 months (baseline) to 6 months, 1 year, 2 years, 3 years, 4 years and 5 years after surgery
  Changes in Forgotten Joint Score (FJS) from 3 months (baseline) to 6 months, 1 year, 2 years, 3 years, 4 years and 5 years after surgery
Survival Rate | 5 years
  Survival rate expressed with Kaplan-Meier estimator at 5 years after surgery
Safety assessment | Intra operative, 3 months, 6 months, 1 year, 3 years, 5 years
  Incidence, type, and severity of all the Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs), and Serious Adverse Device Effects (SADEs) occurred at each follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- The Orthopedic Clinic University Hospital Martin, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: No